CLINICAL TRIAL: NCT00690027
Title: San Diego Bleeding Esophageal Varices Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Marshall J. Orloff, M.D., University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ESTVEPCS
Record Dates: First submitted 2008-06-03; First posted 2008-06-04 (Estimated); Last update posted 2008-06-04 (Estimated); Status verified 2008-06

CONDITIONS: Survival and Control of Bleeding
MeSH Terms: interventions — Emergency Service, Hospital

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Active Comparator): Objective: See Brief Summary, page 2. Eligibility: Patients who require > 2 units blood transfusion for bleeding esophageal varices due to cirrhosis.
  Randomization: By the blind card method to emergency portacaval shunt (EPCS) or emergency endoscopic sclerotherapy (EST) followed by long-term repetitive EST.
  Diagnostic Workup: Completed within 6hr. Rapidity of Therapy: Within 8hr. Failure of Therapy: Bleeding requiring >6u PRBC in first 7 days, or 8 units PRBC during 12 months, or rebleeding after varices were obliterated.
  Rescue Crossover Therapy: When primary therapy has failed. Followup: Lifelong. Data Collection on line, analysis by biostatistician Florin Vaida, PhD External Advisory, Data Monitoring and Safety Committee by 3 senior academicians.
  Interventions: Procedure: Emergency portacaval shunt
- B (Active Comparator): Emergency endoscopic sclerotherapy
  Interventions: Procedure: Emergency and long-term endoscopic sclerotherapy

INTERVENTIONS:
Procedure: Emergency portacaval shunt
  Arms: A
Procedure: Emergency and long-term endoscopic sclerotherapy
  Arms: B

SUMMARY:
In unselected cirrhotic patients with bleeding esophageal varices to compare the influence on mortality rate, duration of life, quality of life, and economic costs of treatment of:

* Emergency portacaval shunt, and
* Emergency and long-term endoscopic sclerotherapy.

DETAILED DESCRIPTION:
See attached Synopsis - APPENDIX 1

ELIGIBILITY:
Inclusion Criteria:

* All patients with UGI bleeding (blood in the esophagus, stomach, or duodenum) who enter the emergency room or develop bleeding while in the hospital or are transferred from nearby hospitals and are suspected of having cirrhosis and BEV will be eligible for consideration (all comers).
* Those who are shown to have the findings of cirrhosis and esophageal varices that:

  * Are seen to be actively bleeding;
  * Have an adherent clot;
  * Have no other associated lesion that could reasonably account for bleeding of that magnitude (such as large gastric or duodenal varices, GU, DU, etc)
* Require 2 or more units of blood transfusion, will be included in the study.

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 211 (Actual)
Dates: Start 1988-04; Primary Completion 1996-08 (Actual); Study Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
Survival | 10 years

SECONDARY OUTCOMES:
Control of bleeding and quality of life | 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Marshall J Orloff, M.D., Principal Investigator — UCSD Medical Center
Locations (1):
- 200 West Arbor Drive, San Diego, California, United States

REFERENCES:
- [Derived] Simonetti RG, Perricone G, Robbins HL, Battula NR, Weickert MO, Sutton R, Khan S. Portosystemic shunts versus endoscopic intervention with or without medical treatment for prevention of rebleeding in people with cirrhosis. Cochrane Database Syst Rev. 2020 Oct 22;10(10):CD000553. doi: 10.1002/14651858.CD000553.pub3. PMID 33089892
- [Derived] Orloff MJ. Fifty-three years' experience with randomized clinical trials of emergency portacaval shunt for bleeding esophageal varices in Cirrhosis: 1958-2011. JAMA Surg. 2014 Feb;149(2):155-69. doi: 10.1001/jamasurg.2013.4045. PMID 24402314
- [Derived] Orloff MJ, Vaida F, Isenberg JI, Wheeler HO, Haynes KS, Jinich-Brook H, Rapier R, Hye RJ, Orloff SL. Child-Turcotte score versus MELD for prognosis in a randomized controlled trial of emergency treatment of bleeding esophageal varices in cirrhosis. J Surg Res. 2012 Nov;178(1):139-46. doi: 10.1016/j.jss.2012.01.004. Epub 2012 Mar 10. PMID 22480831
- [Derived] Orloff MJ, Isenberg JI, Wheeler HO, Haynes KS, Jinich-Brook H, Rapier R, Vaida F, Hye RJ, Orloff SL. A randomized controlled trial of emergency treatment of bleeding esophageal varices in cirrhosis for hepatocellular carcinoma. Am J Surg. 2012 Feb;203(2):182-90. doi: 10.1016/j.amjsurg.2011.02.007. Epub 2011 Jun 16. PMID 21679921
- [Derived] Orloff MJ, Isenberg JI, Wheeler HO, Haynes KS, Jinich-Brook H, Rapier R, Vaida F, Hye RJ. Direct costs of care in a randomized controlled trial of endoscopic sclerotherapy versus emergency portacaval shunt for bleeding esophageal varices in cirrhosis--Part 4. J Gastrointest Surg. 2011 Jan;15(1):38-47. doi: 10.1007/s11605-010-1332-6. Epub 2010 Sep 8. PMID 20824373
- [Derived] Orloff MJ, Isenberg JI, Wheeler HO, Haynes KS, Jinich-Brook H, Rapier R, Vaida F, Hye RJ. Emergency portacaval shunt versus rescue portacaval shunt in a randomized controlled trial of emergency treatment of acutely bleeding esophageal varices in cirrhosis--part 3. J Gastrointest Surg. 2010 Nov;14(11):1782-95. doi: 10.1007/s11605-010-1279-7. Epub 2010 Jul 24. PMID 20658205
- [Derived] Orloff MJ, Isenberg JI, Wheeler HO, Haynes KS, Horacio JB, Rapier R, Vaida F, Hye RJ. Portal-systemic encephalopathy in a randomized controlled trial of endoscopic sclerotherapy versus emergency portacaval shunt treatment of acutely bleeding esophageal varices in cirrhosis. Ann Surg. 2009 Oct;250(4):598-610. doi: 10.1097/SLA.0b013e3181b73126. PMID 19730244
- [Derived] Orloff MJ, Isenberg JI, Wheeler HO, Haynes KS, Jinich-Brook H, Rapier R, Vaida F, Hye RJ. Randomized trial of emergency endoscopic sclerotherapy versus emergency portacaval shunt for acutely bleeding esophageal varices in cirrhosis. J Am Coll Surg. 2009 Jul;209(1):25-40. doi: 10.1016/j.jamcollsurg.2009.02.059. Epub 2009 May 1. PMID 19651060